CLINICAL TRIAL: NCT01661478
Title: Healthcare Provider Attitudes Towards Patients With Substance Use Before and After Implementation of the SBIRT Model in the Emergency Room
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Cheryl McCullumsmith, Division Director, Hospital Psychiatry, University of Alabama at Birmingham
Other Study IDs: X110721008
Record Dates: First submitted 2012-08-07; First posted 2012-08-09 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Patients With Substance Abuse; Healthcare Provider Attitudes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- Emergency Department personnel: survey
  Interventions: Other: Training on motivational interviewing
- Department of Psychiatry personnel: survey
  Interventions: Other: Training on motivational interviewing

INTERVENTIONS:
Other: Training on motivational interviewing

SUMMARY:
The purpose of this quality improvement research project is to briefly survey attitudes among healthcare providers toward patients with substance use disorders before and after substance abuse counselors are placed in the Emergency Room.

DETAILED DESCRIPTION:
The purpose of this quality improvement research project is to briefly survey attitudes among healthcare providers toward patients with substance use disorders before and after substance abuse counselors are placed in the Emergency Room. SBIRT stands for Screening Brief Intervention and Referral to Treatment. The pre-test survey contains 10 questions about attitudes toward patients with substance use disorders and the post-test survey consists of 13 questions about attitudes toward patients with substance use disorders and questions regarding the SBIRT model itself. Health care providers will be surveyed before the SBIRT Counselors begin and again at 6 months, after full SBIRT program with substance counselors on site has been in place, as a part of their regular staff education requirements. Part of the goal of the SBIRT counselors is to educate providers about treatment and analyze data collected by and comments of Emergency Room staff.

ELIGIBILITY:
Inclusion Criteria:

* UAB Emergency Department Staff (attending, resident, nurse, social worker, case manager, patient care technician) or Psychiatry Emergency Services staff (nurses, social workers and residents)

Exclusion Criteria:

* Not employed in UAB Emergency Department

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Personnel in the Emergency Medicine Department and the Department of Psychiatry
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2011-09

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Alabama Birmingham, Birmingham, Alabama